CLINICAL TRIAL: NCT01338831
Title: A Phase I, Multicenter, Open-label Study of LFA102 Administered Intravenously in Patients With Prolactin Receptor-positive Castration-resistant Prostate Cancer or Prolactin Receptor-positive Metastatic Breast Cancer
Brief Title: Phase I Study of LFA102 in Patients With Prolactin Receptor-positive Castration-resistant Prostate Cancer or Prolactin Receptor-positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLFA102X2102; 2011-000494-32 (EudraCT Number)
Record Dates: First submitted 2011-04-14; First posted 2011-04-20 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2017-02

CONDITIONS: Castration-resistant Prostate Cancer; Metastatic Breast Cancer; Uterine Leiomyoma
Keywords: prostate cancer,; breast cancer,; prolactin,; prolactin receptor; uterine leiomyoma
MeSH Terms: conditions — Breast Neoplasms; Myofibroma; Prostatic Neoplasms | interventions — LFA102 monoclonal antibody

ARMS (4):
- Breast & Prostate Cancer Group (Experimental): Dose Escalation
  Interventions: Drug: LFA102
- Breast Cancer Group (Experimental): Dose Expansion
  Interventions: Drug: LFA102
- Prostate Cancer Group (Experimental): Dose Expansion
  Interventions: Drug: LFA102
- Uterine Leiomyoma Group (Experimental): Dose Expansion
  Interventions: Drug: LFA102

INTERVENTIONS:
Drug: LFA102

SUMMARY:
The purpose of this first multi-dose study in cancer patients is to determine the maximum tolerated dose (MTD) or recommended phase II dose (RP2D), characterize the safety, tolerability and pharmacokinetics profile. Once the MTD has been established and/or a RP2D chosen, the study will enroll patients into the expansion portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of prostate cancer, breast cancer, or uterine leiomyoma
2. Detectable metastases by bone scan, CT-scan, or MRI.
3. Presence of prolactin receptor in primary or metastatic tumor (Dose Escalation only)
4. Suitable venous access for blood sampling

Exclusion Criteria:

1. Prior treatment with any anti-prolactin receptor antibody
2. Major surgery within 28 days before study treatment
3. Patients who have received radiotherapy ≤ 2 weeks prior to starting study drug
4. Prior anaphylactic or other severe infusion reaction to antibody formulations

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Incidence rate of Dose Limiting Toxicity | 4 weeks

SECONDARY OUTCOMES:
LFA102 serum concentration | 6 months
Disease response | every 2 to 3 months
Concentrations of antibodies to LFA102 | every month

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (5):
  - Massachusetts General Hospital Mass Gen 3, Boston, Massachusetts
  - Cancer Institute of New Jersey SC, New Brunswick, New Jersey
  - Thomas Jefferson University, Dept. of Phsyciatry & Neurology Thomas Jefferson, Philadelphia, Pennsylvania
  - University of Utah / Huntsman Cancer Institute Huntsman 3, Salt Lake City, Utah
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Modena, MO, Italy
- Novartis Investigative Site, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Agarwal N, Machiels JP, Suarez C, Lewis N, Higgins M, Wisinski K, Awada A, Maur M, Stein M, Hwang A, Mosher R, Wasserman E, Wu G, Zhang H, Zieba R, Elmeliegy M. Phase I Study of the Prolactin Receptor Antagonist LFA102 in Metastatic Breast and Castration-Resistant Prostate Cancer. Oncologist. 2016 May;21(5):535-6. doi: 10.1634/theoncologist.2015-0502. Epub 2016 Apr 18. PMID 27091421
- See also: Results for CLFA102X2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13004